CLINICAL TRIAL: NCT04479267
Title: A Phase II Study Evaluating Safety and Efficacy of Polatuzumab Vedotin in Combination With Rituximab, Cyclophosphamide, Doxorubicin, and Prednisone in Patients With Previously Untreated Double and Triple Hit Lymphoma, Double Expressor Lymphoma and High-Grade B Cell Lymphoma
Brief Title: Polatuzumab Vedotin and Combination Chemotherapy for the Treatment of Previously Untreated Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Dipenkumar Modi, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-135; P30CA022453 (NIH)
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Diffuse Large B-Cell Lymphoma; High Grade B-Cell Lymphoma w/MYC & BCL2 or BCL6 Rearrangements; High Grade B-Cell Lymphoma w/MYC, BCL2 & BCL6 Rearrangements; Double Expressor Lymphoma; High-grade B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Prednisone; Prednisolone; Methylprednisolone; exifone; Rituximab; CT-P10; polatuzumab vedotin; Cyclophosphamide; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (polatuzumab vedotin, R-CHP) (Experimental): Patients receive prednisone PO, prednisolone IV, or methylprednisolone IV on days 1-5. Patients also receive rituximab IV, polatuzumab vedotin IV over 30-90 minutes, cyclophosphamide IV, and doxorubicin hydrochloride IV on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Prednisone; Drug: Prednisolone; Drug: Methylprednisolone; Biological: Rituximab; Drug: Polatuzumab Vedotin; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride

INTERVENTIONS:
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone, 1, 2-Dehydrocortisone, 17,21-Dihydroxypregna-1,4-diene-3,11,20-trione, 53-03-2, Adasone, Cortancyl, Dacortin, , Decortisyl, Decorton, Delta 1-Cortisone, Delta-Dome
Drug: Prednisolone — Given IV
  Other Names: (11beta)-11,17,21-Trihydroxypregna-1,4-diene-3,20-dione, .delta.1-Hydrocortisone, 1,2-Dehydrohydrocortisone, 50-24-8, 9120, Adnisolone, Aprednislon, Capsoid, Cortalone, Cortisolone
Drug: Methylprednisolone — Given IV
  Other Names: (6alpha,11beta)-11,17,21-Trihydroxy-6-methylpregna-1,4-diene-3,20-dione, 6Alpha-Methylprednisolone, Adlone, Caberdelta M, DepMedalone, Depo Moderin, Depo-Nisolone, Duralone, Emmetipi, Esametone
Biological: Rituximab — Given IV
  Other Names: 174722-31-7, 687451, ABP 798, BI 695500, C2B8 Monoclonal Antibody, Chimeric Anti-CD20 Antibody, CT-P10, IDEC-102, IDEC-C2B8, IDEC-C2B8 Monoclonal Antibody, MabThera, Monoclonal Antibody IDEC-C2B8
Drug: Polatuzumab Vedotin — Given IV
  Other Names: 1313206-42-6, ADC DCDS4501A, Antibody-Drug Conjugate DCDS4501A, DCDS4501A, FCU 2711, POLATUZUMAB VEDOTIN, polatuzumab vedotin-piiq, Polivy, RG7596, Ro 5541077-000
Drug: Cyclophosphamide — Given IV
  Other Names: 1-bis(2-chloroethyl)-amino-1-oxo-2-aza-5-oxaphosphoridin monohydrate, 2-[bis(2-chloroethyl)amino]tetrahydro-2H-1,3,2-oxazaphosphorine 2-oxide monohydrate
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 14-Hydroxydaunorubicin Hydrochloride, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-

SUMMARY:
This phase II trial studies how well polatuzumab vedotin and combination chemotherapy work in treating patients with previously untreated double, triple hit lymphoma, Double Expressor Lymphoma or High-Grade B Cell Lymphoma. Polatuzumab vedotin is a monoclonal antibody that works by binding with cancer cells and releasing another chemotherapy drug, called monomethyl auristatin E, into the cell causing the cancer cells to die or stop growing. Chemotherapy drugs, such as rituximab, cyclophosphamide, doxorubicin, and prednisone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving polatuzumab vedotin with combination chemotherapy may work better in treating patients with double or triple hit lymphoma compared to combination chemotherapy alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the rate of complete remission (CR) with polatuzumab vedotin plus rituximab, cyclophosphamide, doxorubicin hydrochloride, and prednisone (R-CHP) in patients with newly diagnosed previously untreated double, triple hit lymphoma, Double Expressor Lymphoma or High-Grade B Cell Lymphoma. as measured by positron emission tomography (PET)-defined CR rate using the modified Lugano response criteria at the time of primary response assessment (6-8 weeks after cycle 6 day 1 or last dose of study medication).

PRIMARY OBJECTIVE:

I. To determine the rate of complete remission (CR) with polatuzumab vedotin plus rituximab, cyclophosphamide, doxorubicin hydrochloride, and prednisone (R-CHP) in patients with newly diagnosed previously untreated double, triple hit lymphoma, Double Expressor Lymphoma or High-Grade B Cell Lymphoma. as measured by positron emission tomography (PET)-defined CR rate using the modified Lugano response criteria at the time of primary response assessment (6-8 weeks after cycle 6 day 1 or last dose of study medication).

SECONDARY SAFETY OBJECTIVE:

I. To evaluate the safety and tolerability of the combination of polatuzumab vedotin (PoV) plus R-CHP as defined by Common Terminology Criteria for Adverse Events (CTCAE) 5.0.

SECONDARY EFFICACY OBJECTIVES:

I. To assess the progression free survival (PFS) with PoV plus R-CHP in the above-mentioned patient population.

II. To assess the overall survival (OS) with PoV plus R-CHP in the above-mentioned patient population.

III. To assess the overall response rate (ORR; complete response [CR] or partial response [PR]) at the time of primary response assessment, based on modified Lugano PET-computed tomography (CT) criteria, as determined by the investigator.

IV. To assess the duration of response (DOR) to PoV plus R-CHP based on PET-CT, as determined by the investigators in the above-mentioned patient population.

EXPLORATORY OBJECTIVES:

I. To explore the relationship between CD79b expression and response to treatment with PoV plus R-CHP.

II. To explore the relationship between MYC expression and response to treatment with PoV plus R-CHP.

III. To explore polatuzumab vedotin treatment on Myc protein expression.

OUTLINE:

Patients receive prednisone orally (PO), prednisolone intravenously (IV), or methylprednisolone IV on days 1-5. Patients also receive rituximab IV, polatuzumab vedotin IV over 30-90 minutes, cyclophosphamide IV, and doxorubicin hydrochloride IV on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF)
* Previously untreated patients (except for one prior cycle of CHOP+R) with diffuse large B-cell lymphoma (DLBCL) as determined by local pathology. World Health Organization (WHO) histologies will include:

  * Double hit lymphoma (DHL) or triple hit lymphoma (THL) confirmed by fluorescence in situ hybridization (FISH) testing by local pathology (defined as MYC and BCL2 and/or BCL6 rearrangements)
  * High grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements
  * Double expressor lymphoma (DEL) defined as overexpression of MYC(> or = to 40%) and BCL2 (> or = to 50%) identified by immunohistochemistry (IHC)
  * High grade B-cell lymphoma (HGBL) NOS subtype
* Availability of archival formalin-fixed paraffin-embedded (FFPE) tissue blocks or 15 unstained slides serial sections (3-5 um in thickness) prior to study enrollment. The pathology report must be available for review and a tissue block sent for retrospective central confirmation of diagnosis. If central confirmation is unable to be performed on submitted material, stained slides used for diagnosis and/or additional tumor tissue specimens may also be requested

  * For clarification: Only availability of tumor sample must be verified prior to C1D1 however treatment can commence prior to completion of central review. The adequacy of the tissue will be confirmed if possible (ie. if it will not delay treatment).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Life expectancy of at least 24 weeks
* At least one bi-dimensionally measurable lesion > 1.5 cm in its longest dimension as measured by CT or magnetic resonance imaging (MRI)
* Ability and willingness to comply with the study protocol procedures
* Left ventricular ejection fraction (LVEF) >= 45% on cardiac multiple-gated acquisition (MUGA) scan or cardiac echocardiogram (ECHO)
* Hemoglobin >= 8.0 g/dL without packed RBC transfusion during 14 days before first treatment (unless due to underlying disease, as established by extensive bone marrow involvement or due to hypersplenism secondary to the involvement of the spleen by DLBCL per the investigator)
* Absolute neutrophil count (ANC) >= 1,000/uL (unless due to underlying disease, as established by extensive bone marrow involvement or due to hypersplenism secondary to the involvement of the spleen by DLBCL per the investigator)
* Platelet count >= 75,000/uL (unless due to underlying disease, as established by extensive bone marrow involvement or due to hypersplenism secondary to the involvement of the spleen by DLBCL per the investigator)
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 12 months after the last dose of study treatment

  * A woman is considered to be of childbearing potential if she is post-menarcheal, has not reached a postmenopausal state (>= 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus)
  * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices
  * Women must refrain from donating eggs during the same period
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception
* For women of childbearing potential, a negative serum pregnancy test result within 7 days prior to commencement of dosing. Women who are considered not to be of childbearing potential are not required to have a pregnancy test
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below:

  * With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 5 months after the last dose of polatuzumab vedotin, 3 months after the last dose of rituximab, and for at least 6 months after the last dose of cyclophosphamide to avoid exposing the embryo for the duration of the pregnancy. Men must refrain from donating sperm during this same period
* Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception. Male patients considering preservation of fertility should bank sperm before study treatment
* CRITERIA FOR TISSUE SUBMISSION:
* Eligible patients must have available at the study site a representative formalin-fixed, paraffin-embedded tumor specimen that enabled the definitive diagnosis of DLBCL

  * The specimen must contain adequate evaluable tumor cells (>= 20% for excisional biopsy and >= 50% if sample is a core biopsy) to enable relevant biomarker analysis
  * A tissue block (preferred) or 15 serial, freshly cut, unstained slides plus punch biopsy of the tissue block accompanied by an associated pathology report will be requested. Punch biopsy is required only with the slide submission. Cytological or fine-needle aspiration samples are not acceptable
  * If the archival tissue is unavailable or insufficient on the basis of the above criteria, the patient may still be eligible if the patient is willing to provide tissue from a pretreatment core or excisional/incisional biopsy of the tumor. Cytological or fine-needle aspiration samples are not acceptable. The sample should be shipped according to instructions provided in the laboratory manual. Tissue collected on study will not be returned to sites. If needed, additional slides from previously collected samples may be requested. Cases received from each of the participating institutes should be histological confirmed according to the 2016 WHO classification of tumors of hematopoietic and lymphoid neoplasm. The evaluation process by immunohistochemistry (IHC) and fluorescent in situ hybridization (FISH) requires the possession of representative amount of tissues in a paraffin embedded block to be sent to the primary testing institution (Karmanos Cancer Center, Detroit, Michigan). Shipped slides should be placed in proper containers to avoid breakage during shipping. Blocks of paraffin embedded tissue or slides should be sent with a tracking number the address. In addition, the participation institution should call the laboratory at 313-576-8351 (Julie Boerner) for any sample that they ship and provide tracking number

Exclusion Criteria:

* Contraindication to any of the individual components of R-cyclophosphamide, doxorubicin hydrochloride, oxaliplatin, prednisone (CHOP) or any component of PoV, including prior receipt of anthracyclines or history of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies (MAbs) (or recombinant antibody-related fusion proteins) or known sensitivity or allergy to murine products
* Contraindication to rituximab or prior administration of an anti CD 20 antibody
* Treatment with radiotherapy, chemotherapy, immunotherapy, immunosuppressive therapy, or any investigational agent for the purposes of treating cancer prior to cycle 1 day 1 with the following exceptions:

  * One prior treatment cycle of CHOP+R is allowed. Patients who received one prior R-CHOP will receive 6 cycles of R-CHP plus Polatuzumab Vedotin per protocol treatment.
  * Glucocorticoid treatment required for lymphoma symptom control prior to the start of study treatment, prednisone 100 mg or equivalent can be given for a maximum of 13 days as a prephase treatment, with all tumor assessments completed prior to starting prednisone
  * One dose of prophylactic intrathecal chemotherapy with methotrexate
* Grade 3b follicular lymphoma
* Primary mediastinal (thymic) large B-cell lymphoma
* Burkitt lymphoma
* Primary or secondary central nervous system (CNS) lymphoma (primary or secondary involvement), primary effusion DLBCL, and primary cutaneous DLBCL
* Current grade 2 peripheral neuropathy per Common Terminology Criteria for Adverse Events (CTCAE) 5.0
* History of other malignancy that could affect compliance with the protocol or interpretation of results. Exceptions include, but are not limited to:

  * Patients with a history of curatively treated basal or squamous cell carcinoma of the skin, in situ carcinoma of the cervix or ductal carcinoma in situ of the breast at any time prior to the study are eligible
  * A patient with any other malignancy that has been treated with surgery alone with curative intent and the malignancy has been in remission without treatment for >= 3 years prior to enrollment is eligible
  * Patients with low-grade, early-stage prostate cancer with no requirement for therapy at any time prior to study are eligible
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results, including significant cardiovascular disease (such as New York Heart Association class III or IV cardiac disease, myocardial infarction within the last 6 months, unstable arrhythmias, or unstable angina) or significant pulmonary disease (including obstructive pulmonary disease and history of bronchospasm)
* History or presence of an abnormal electrocardiogram (ECG) that is clinically significant in the investigator's opinion, including complete left bundle branch block, second- or third-degree heart block
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment or any major episode of infection requiring treatment with intravenous (IV) antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks prior to cycle 1 day 1
* Patients with clinical suspicion of active or latent tuberculosis (to be confirmed by a positive interferon gamma release assay)
* Positive test results for chronic hepatitis B virus (HBV) infection (defined as positive hepatitis B surface antigen [HBsAg] serology)

  * Patients with occult or prior HBV infection (defined as negative HBsAg and positive hepatitis B core antibody [HBcAb]) may be included if HBV deoxyribonucleic acid (DNA) polymerase chain reaction (PCR) is undetectable, provided that they are willing to undergo DNA testing on day 1 of every cycle and monthly for at least 12 months after the last cycle of study treatment. Patients who have protective titers of hepatitis B surface antibody (HBsAb) after vaccination or prior but cured hepatitis B are eligible
* Positive test results for hepatitis C virus (HCV) antibody

  * Patients who are positive for HCV antibody are eligible only if PCR is negative for HCV ribonucleic acid (RNA)
* Known history of human immunodeficiency virus (HIV) seropositive status

  * For patients with unknown HIV status, HIV testing will be performed at screening
* Vaccination with a live vaccine within 28 days prior to treatment
* Recent major surgery (within 6 weeks before the start of cycle 1 day 1) other than for diagnosis
* Women who are pregnant or lactating or who intend to become pregnant within a year of the last dose of study treatment
* Patients with a history of progressive multifocal leukoencephalopathy
* Creatinine > 1.5 x ULN or a measured creatinine clearance < 40 mL/min (unless abnormal laboratory values are due to underlying lymphoma per the investigator)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 x ULN (unless abnormal laboratory values are due to underlying lymphoma per the investigator)
* Total bilirubin >= 1.5 x ULN (unless abnormal laboratory values are due to underlying lymphoma per the investigator)

  * Patients with documented Gilbert disease may be enrolled if total bilirubin is =< 3 x ULN
* International normalized ratio (INR) or prothrombin time (PT) > 1.5 x ULN in the absence of therapeutic anticoagulation (unless abnormal laboratory values are due to underlying lymphoma per the investigator)
* Partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) > 1.5 x ULN in the absence of a lupus anticoagulant (unless abnormal laboratory values are due to underlying lymphoma per the investigator)
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* The use of Evushield or other post-exposure anti-viral medications against COVID19 does not affect study eligibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2026-07-19 (Estimated)

PRIMARY OUTCOMES:
Rate of complete remission | Up to 6-8 weeks after cycle 6 day 1 (cycles = 21 days) or last dose of study medication
  Will be assessed by modified Lugano response criteria for malignant lymphoma. The complete remission rate will be summarized by a binomial response rate and its associated 2-sided 80% confidence interval (CI) using Pearson-Klopper method. The primary efficacy analysis will be also performed based on all response evaluable subjects as a sensitivity analysis.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 30 days after last dose of study treatment
  Safety will be assessed through summaries of adverse events, summaries of changes from screening assessments in laboratory test results, electrocardiograms, and changes in vital signs. All adverse events occurring on or after first study treatment will be summarized by mapped term, appropriate thesaurus levels, and National Cancer Institute (NCI) Common Terminology Criteria Adverse Events version (v) 4.03 toxicity grade. All serious adverse events will be listed separately and summarized. Deaths reported during the study treatment period and those reported during follow-up after treatment discontinuation will be listed. Relevant laboratory and vital sign (temperature, heart rate, respiratory rate, pulse oximetry, and blood pressure) data will be displayed by time, with NCI Common Terminology Criteria for Adverse Events v5.0. Grade 3 and 4 values identified where appropriate.
Progression-free survival (PFS) | From the start date of the treatment until the date of progression or death from any cause, whichever occurs first, assessed up to 12 months
  The distribution of PFS will be graphically summarized using the Kaplan-Meier (KM) curve and the median PFS and its associated 2-sided CI will be estimated using the KM estimator. The median follow-up time and its 2-sided CI will be estimated using the reverse KM estimator.
Overall response rate (ORR) | Up to 12 months
  Will be defined as complete response (CR) or partial response (PR) at primary response assessment based on positron emission tomography/computed tomography as determined by the investigator and assessed using modified Lugano response criteria. CR and PR will be summarized using frequency and percentage. The ORR will be summarized by a binomial response rate and its associated 2-sided CI using Pearson-Klopper method.
Duration of response (DOR) | From the date of CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is documented among all treated subjects who had a confirmed CR or PR, assessed up to 12 months
  The distribution of DOR will be graphically summarized using the KM curve and the median PFS and its associated 2-sided CI will be estimated using the KM estimator.

OTHER OUTCOMES:
Biomarker assessment | Up to time of disease progression, assessed up to 12 months
  Exploratory analyses of biomarkers related to tumor biology and the mechanisms of action of polatuzumab vedotin and rituximab will be conducted. Analyses will assess prognostic and/or predictive value of candidate biomarkers separately for each histological subtype and both investigator and Independent Review Committee assessed outcomes. Specifically, the association between candidate biomarkers and positron emission tomography (PET)-computed tomography (CT) CR rate and objective response rate and potentially other measures of efficacy and safety, independent of treatment, will be explored to assess potential prognostic value. In addition, the potential effect modification of treatment effect on PET-CT CR rate and OR rate and potentially other measures of efficacy and safety, by biomarker status, will be explored to assess potential predictive value.

CONTACTS AND LOCATIONS:
Overall Officials: Dipenkumar Modi, M.D., Principal Investigator — Barbara Ann Karmanos Institute
Locations (1):
- Karmanos Cancer Institute, Detroit, Michigan, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-04): https://cdn.clinicaltrials.gov/large-docs/67/NCT04479267/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT04479267/ICF_001.pdf